CLINICAL TRIAL: NCT04694482
Title: The Psychopathological Impact of the SARS-CoV-2 Epidemic on Subjects Suffering From Mental Disorders: Data From ASST Monza
Brief Title: The Impact of the COVID-19 (SARS-CoV-2 Disease) on Psychopathology
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Fabrizia Colmegna, Medical Doctor, University of Milano Bicocca
Other Study IDs: COVID-19-psychiatry
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2022-10

CONDITIONS: Psychosis;Schizophrenic; Personality Disorders; Mood Disorders; Anxiety Disorders; Post Traumatic Stress Disorder
MeSH Terms: conditions — Personality Disorders; Mood Disorders; Anxiety Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psychiatric patients: Psychometric scales
  Interventions: Other: Psychometric scale administration
- healthy controls: Psychometric scales
  Interventions: Other: Psychometric scale administration

INTERVENTIONS:
Other: Psychometric scale administration — PTSD symptoms are assessed using a specific scale (IES-R) and compared between the two groups

SUMMARY:
The outbreak of the SARS-CoV-2 pandemic may be considered a traumatic phenomenon.

In a sample of subjects suffering from different psychiatric disorders, psychopathological status and Post-Traumatic Stress Disorder (PTSD) symptoms over time are assessed using specific psychometric scales. In a sample of healthy controls PTSD symptoms are evaluated by Impact of Event Scale Revised (IES-R) and compared to patients' scores.

We hypothesize that a significant number of psychiatric outpatients have experienced a clinical psychopathological worsening and a greater prevalence of PTSD symptoms compared to the general population. The study of the potential psychopathological changes could represent a useful contribution to deepen the understanding of psychological consequences of the pandemic.

DETAILED DESCRIPTION:
SARS-CoV-2 epidemic is a worldwide phenomenon which generated fear, anxiety, depression and PTSD symptoms, as a consequence of the high number of deaths and the restricted measures adopted by the Italian Government to stem the spread of the virus.

The aims of the study are: (1) to investigate potential psychopathological changes over time in a sample of patients affected by different psychiatric disorders (schizophrenia, bipolar disorder, major depression, anxiety/Obsessive-Compulsive Disorder (OCD), personality disorders); (2) to compare patients and healthy controls in terms of post-traumatic symptoms.

Outpatients affected by different psychiatric disorders are recruited during their routine visits and demographic/clinical variables are collected from their medical records.

Psychopathological status and PTSD symptoms are retrospectively assessed using specific psychometric scales, such as Brief Psychiatry Rating Scale (BPRS), Clinical Global Impression (CGI), Disability Scale (DISS), Hamilton Anxiety Rating Scale (HAM-A), Hamilton Depression Rating Scale (HAM-D), Montgomery and Asberg Depression Rating Scale (MADRS), Young Mania Rating Scale (YMRS), Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), IES-R.

The assessment is performed over time at three time points: T0 corresponding to the outbreak of the pandemic (January-February 2020), T1 which was the lockdown period (March-April 2020) and T2 corresponding to the reopening and restarting (May-June 2020).

Descriptive analyses of the whole sample will be performed. Then, mixed linear regression models will be run to investigate the change over time in patients' psychometric scores and whether it differs among different diagnostic groups. Moreover, same analyses will be performed to compare patients and healthy subjects in terms of change of IES-R scores over time.

ELIGIBILITY:
Inclusion Criteria:

* understanding of the Italian language
* ability to understand and sign written informed consent

Exclusion Criteria:

* severe mental retardation
* pregnancy or post-partum period
* severe or chronic medical condition
* health workers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychiatric outpatients and healthy controls resident in the same geographic area as the patients
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizia Colmegna, MD, Principal Investigator — ASST Monza
Locations (1):
- University of Milan Bicocca - Ospedale San Gerardo, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tagliabue I, Caldiroli A, Capuzzi E, Borgonovo R, Scalia A, Ferre A, Sibilla M, Turco M, Affaticati LM, Crespi G, Galimberti G, Dakanalis A, Colmegna F, Buoli M, Clerici M. Which Factors Are Associated With Comorbid Psychiatric Conditions in Patients Affected by Substance Use Disorders? The Impact of COVID-19 Pandemic on Dual-Diagnosis Subjects. J Dual Diagn. 2024 Jul-Sep;20(3):201-209. doi: 10.1080/15504263.2024.2346519. Epub 2024 May 10. PMID 38728603
- [Derived] Caldiroli A, Tagliabue I, Turco M, Capuzzi E, Fortunato A, Tringali A, Montana C, Maggioni L, Pellicioli C, Sibilla M, Marcatili M, Crespi G, Colmegna F, Buoli M, Clerici M. Comparing the COVID-19-related PTSD symptoms between psychiatric patients and healthy subjects: an observational retrospective study from Northern Italy. Psychol Health Med. 2023 Jun;28(5):1298-1308. doi: 10.1080/13548506.2022.2121971. Epub 2022 Sep 11. PMID 36093977
- [Derived] Caldiroli A, Capuzzi E, Tringali A, Tagliabue I, Turco M, Fortunato A, Sibilla M, Montana C, Maggioni L, Pellicioli C, Marcatili M, Nava R, Crespi G, Colmegna F, Buoli M, Clerici M. The psychopathological impact of the SARS-CoV-2 epidemic on subjects suffering from different mental disorders: An observational retrospective study. Psychiatry Res. 2022 Jan;307:114334. doi: 10.1016/j.psychres.2021.114334. Epub 2021 Dec 7. PMID 34902818

RESULTS

PARTICIPANT FLOW:
Groups:
- Psychiatric Patients: Patients with different psychiatric diagnoses are included. All the psychometric scales are administered.
  PTSD symptoms are assessed using a specific scale (IES-R) and compared with healthy controls
- Healthy Controls: PTSD symptoms are assessed using a specific scale (IES-R) and compared with psychiatric patients.
Period: Overall Study
Arm/Group | Psychiatric Patients | Healthy Controls
Started | 200 | 70
Completed | 166 | 57
Not Completed | 34 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychiatric Patients | Healthy Controls | Total
Number analyzed (Participants) | 166 | 57 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.22 (14.23) | 43.86 (15.19) | 47.85 (14.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 32 | 111
  Male | 87 | 25 | 112
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 166 | 57 | 223
Education [Count of Participants; unit: Participants]
  Primary school | 11 | 0 | 11
  Secondary school | 69 | 2 | 71
  High school | 77 | 15 | 92
  Graduate | 9 | 28 | 37
  Post-graduate | 0 | 12 | 12
Marital status [Count of Participants; unit: Participants]
  Single | 92 | 13 | 105
  Married/cohabitant | 46 | 40 | 86
  Separated/divorced | 23 | 2 | 25
  Widower | 5 | 2 | 7
Occupational status [Count of Participants; unit: Participants]
  Employed | 45 | 45 | 90
  Unemployed | 27 | 5 | 32
  Never-before-employed | 3 | 0 | 3
  Invalid-at-work | 75 | 0 | 75
  Retired | 16 | 7 | 23
Family history of psychiatric disorders [Count of Participants; unit: Participants]
  None | 81 | 44 | 125
  Schizophrenia | 19 | 2 | 21
  Bipolar Disorder | 6 | 0 | 6
  Major Depressive Disorder | 33 | 10 | 43
  Anxiety disorders | 13 | 0 | 13
  Eating disorder | 2 | 0 | 2
  Drug abuse | 6 | 1 | 7
  Personality Disorders | 6 | 0 | 6
Substance abuse [Count of Participants; unit: Participants]
  None | 119 | 49 | 168
  Alcohol | 15 | 0 | 15
  Cannabis | 17 | 7 | 24
  Cocaine | 8 | 0 | 8
  Heroin | 4 | 0 | 4
  Benzodiazepines | 1 | 1 | 2
  Gambling | 2 | 0 | 2
Medical comorbility [Count of Participants; unit: Participants]
  Yes | 86 | 12 | 98
  No | 80 | 45 | 125
6-months pre-COVID poly-abuse [Count of Participants; unit: Participants]
  Yes | 18 | 0 | 18
  No | 148 | 57 | 205
6-months post-COVID poly-abuse [Count of Participants; unit: Participants]
  Yes | 8 | 0 | 8
  No | 158 | 57 | 215
Presence of 2 COVID symptoms [Count of Participants; unit: Participants]
  Yes | 5 | 20 | 25
  No | 161 | 37 | 198
Medical poly-comorbility [Count of Participants; unit: Participants]
  Yes | 57 | 4 | 61
  No | 109 | 53 | 162

OUTCOME MEASURES:

1. Primary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: Range 0-126. Higher scores mean worse outcome. This psychometric scale measures the global psychopathology investigating several psychopathological areas (anxiety, thinking, mood, perception, etc.). It provides a global score of severity (> 31 means that the patient need hospitalization).
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only psychiatric patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 166
score on a scale
  T0 | 29.30 (10.41)
  T1 | 32.80 (11.04)
  T2 | 30.25 (9.4)

2. Primary Outcome: Clinical Global Impression (CGI) Severity Subscale
Description: Range 0-7. Higher scores mean worse outcome. The severity subscale measures the global severity of symptom presentation based on the clinicians' evaluation (Normal, Borderline mentally ill, Mildly ill, etc.).
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only psychiatric patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 166
score on a scale
  T0 | 4.02 (1.31)
  T1 | 4.23 (1.29)
  T2 | 4.10 (1.31)

3. Primary Outcome: Clinical Global Impression (CGI) Improvement Subscale
Description: Range 0-7. Higher scores mean worse outcome. The improvement subscale measures the clinical improvement (how much has the patient changed) according to the clinician's judgement. It results as: very much improved, much improved, minimally improved, no changed, minimally worse, etc.).
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only psychiatric patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 166
score on a scale
  T1 | 4.37 (0.97)
  T2 | 3.61 (0.91)

4. Primary Outcome: Hamilton Anxiety Scale (HAM-A)
Description: Range 0-56. Higher scores mean worse outcome. The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety).
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only psychiatric patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 166
score on a scale
  T0 | 6.81 (8.13)
  T1 | 10.03 (9.02)
  T2 | 7.92 (8.71)

5. Primary Outcome: Impact of Event Scale - Revised Version (IES-R)
Description: Range 0-88. Higher scores mean worse outcome. The scale is a self-report measure of current subjective distress in response to a specific traumatic event. It comprises 3 subscales representative of the major symptom clusters of post-traumatic stress: intrusion, avoidance, and hyper-arousal.
Time Frame: 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Both psychiatric patients and healthy controls were assessed for this outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients | Healthy Controls
Number analyzed (Participants) | 166 | 57
score on a scale
  T1 | 20.18 (18.29) | 24.34 (12.91)
  T2 | 13.47 (15.15) | 20.57 (13.37)

6. Secondary Outcome: Disability Scale (DISS)
Description: Range 0-30. Higher scores mean worse outcome. The scale includes 3 self-rated items designed to measure the extent to which 3 major domains (work 0-10, social life/leisure activities 0-10, and family life/home responsibilities 0-10) in the patient's life are functionally impaired by psychiatric or medical symptoms. For each subscale, higher scores mean better outcome. Subscales are summed to compute a total score.
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only psychiatric patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 166
score on a scale
  T0 | 17.95 (7.90)
  T1 | 17.50 (7.57)
  T2 | 17.25 (8.01)

7. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D)
Description: Range 0-67. Higher scores mean worse outcome. The scale measures the severity of depressive symptoms taking into account anxiety and somatic manifestations.
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only bipolar and major depressed patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 65
score on a scale
  T0 | 7.42 (6.44)
  T1 | 12.57 (12.45)
  T2 | 8.03 (6.90)

8. Secondary Outcome: Montgomery and Asberg Depression Rating Scale (MADRS)
Description: Range 0-60. Higher scores mean worse outcome. The scale measures the core symptoms of depression (e.g. anhedonia).
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only bipolar and major depressed patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 65
score on a scale
  T0 | 9.45 (8.52)
  T1 | 12.91 (9.52)
  T2 | 9.69 (8.32)

9. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: Range 0-56. Higher scores mean worse outcome. The scale has 11 items and is based on the patient's subjective report of his or her clinical condition, and generally limited to the previous 48 hours. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale.
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only bipolar patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 29
score on a scale
  T0 | 3.14 (5.84)
  T1 | 4.69 (9.04)
  T2 | 3.51 (7.04)

10. Secondary Outcome: Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)
Description: Range 0-40. Higher scores mean worse outcome. The scale is a semi-structured interview that consists of 10 core items, 5 measuring time, interference, distress, resistance and control of obsessions (items: 1-5), and 5 identical items measuring compulsions (items: 6-10). The items are rated from 0 (no symptoms) to 4 (severe symptoms), and yield a global severity score (range 0-40).
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only Obsessive-Compulsive patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 7
score on a scale
  T0 | 9.20 (10.00)
  T1 | 10.40 (10.87)
  T2 | 10.20 (11.49)

11. Secondary Outcome: Positive And Negative Syndrome Scale (PANSS)
Description: Range 30-210. Higher scores mean worse outcome. The scale is a medical scale used for measuring symptom severity of patients with schizophrenia. It assesses positive symptoms, which refer to an excess or distortion of normal functions (e.g., hallucinations and delusions), and negative symptoms, which represent a diminution or loss of normal functions. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers.
Time Frame: 2 months at the start of outbreak (T0), 2 months of lockdown period (T1) and 2 months of reopening phase (T2)
Population: Only Schizophrenia patients were assessed for this outcome; data not collected for healthy controls.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychiatric Patients
Number analyzed (Participants) | 66
score on a scale
  T0 | 60.72 (27.33)
  T1 | 62.49 (32.96)
  T2 | 62.63 (25.85)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed. We did not test any new compound in the study. The causes of mortality are the same as those of the general population
Arm/Group | Psychiatric Patients | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT04694482/Prot_SAP_000.pdf